CLINICAL TRIAL: NCT06105944
Title: Economic Evaluation of Lower Limb Prostheses in the Netherlands Including the Cost-effectiveness of Non-microprocessor Controlled Knees Versus Microprocessor Controlled Knees
Brief Title: Economic Evaluation of Lower Limb Prostheses for Persons With a Knee-disarticulation or Transfemoral Amputation
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 671860-cost
Record Dates: First submitted 2023-08-23; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Amputation; Prosthesis User; Prosthesis
Keywords: cost-effectiveness; microprocessor knee; economic evaluation; transfemoral amputation; knee-disarticulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective questionnaire study is to evaluate the cost-effectiveness of non-microprocessor controlled prosthetic knees (NMPK) versus microprocessor controlled prosthetic knees (MPK) in persons with a knee-disarticulation or transfemoral amputation. The main aims are:

* to provide an overview of the costs, health-related quality of life, and user experiences associated with the use of different types of prosthetic knees.
* to evaluate the cost-effectiveness of the NMPK compared to the MPK for adult prosthesis users.

Participants will fill out three questionnaires about (1) their medical consumption and productivity costs; (2) health-related quality of life; (3) utility, ambulation and well-being.

Researchers will compare the persons with a NMPK to the persons with an MPK to investigate the cost-efficiency of both types of knees.

DETAILED DESCRIPTION:
A transfemoral amputation or knee disarticulation can have a negative influence on a person's daily activities, participation, and other aspects of daily life. In previous studies it has been suggested that the use of a microprocessor-controlled knee (MPK) can help increase functional mobility, decrease falls and stumbles and improve quality of life. Although there is a hefty cost associated with this type of knee, it is not certain this outweighs the potential gains.

ELIGIBILITY:
Inclusion Criteria:

* At least one year post amputation
* Able to read and write in Dutch
* Use a prosthesis with socket

Exclusion Criteria:

* Bilateral amputation
* Osseointegration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults with a unilateral knee-disarticulation or transfemoral amputation who use a prosthesis with an NMPK or MPK.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2022-12-17 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Costs related to lower limb prosthesis use | At the baseline, participants were asked to fill out the questionnaire over a retrospective period of six months
  To get insight in the costs, two existing questionnaires were combined: the Productivity Cost Questionnaire (iPCQ) and the Medical Consumption Questionnaire (iMCQ).
  The iMCQ is used to measure medical consumption. It includes questions related to the number of appointments with health care providers. The iPCQ measures and values productivity losses. It looks at absenteeism, presenteeism, productivity losses and unpaid work. As this study focussed on costs related to lower limb prostheses, questions about appointments with a dietician and speech therapist, and trips to the emergency room were replaced with questions about the type of prosthesis and the number of appointments with their prosthetist. Finally, questions about personal costs related to the acquisition and repairs of the prosthesis, as well as personal expenses were added. As this questionnaire looks at number of appointments and costs, there is no minimum or maximum value score.
Health-related quality of life (HRQOL) 1 | At the baseline, participants were asked to fill out the questionnaire based on their health status that day.
  To evaluate the HRQOL, participants were asked to fill out the Dutch version of the EuroQol - five dimensions - five levels (EQ-5D-5L). This is a self-assessment tool that consists of five questions about mobility, self-care, daily activities, pain and anxiety/depression. For each question, the participant can answer with five response levels: no problems, slight problems, moderate problems, severe problems, extreme problems/unable to do so. The Dutch scoring algorithm for the EQ-5D-5L was used to compute a solitary value representing the health status of the participant. The calculated values fall within the range of -0.446 to 1, where higher scores denote enhanced HRQOL.
Health-related quality of life (HRQOL) 2 | At the baseline, participants were asked to fill out the questionnaire based on their health status that day.
  At the end of the EQ-5D-5L, participants were asked to rate their perceived health that day on a visual analogue scale (VAS) of 0 (worst health imaginable) to 100 (best health imaginable).
Prosthesis-related quality of life | At the baseline, participants were asked to fill out the questionnaire over a retrospective period of four weeks.
  To measure the prosthesis related quality of life, participants filled out parts of the Prosthesis Evaluation Questionnaire (PEQ). The PEQ is a self-report questionnaire to evaluate prosthesis and prosthesis-related quality of life. Questions focus on use, satisfaction, quality of life, tripping and falling. The subscales used in the PEQ are not dependent on each other and can therefore be used independently to fit the research question. For this study, three subscales were utilized: utility, ambulation and well-being.
  The questions are scored on a visual analogue scale (VAS) from 0-100. A higher score on this questionnaire is linked to a more positive outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Livit Orthopedie, Amsterdam
  - OIM Orthopedie, Assen

IPD SHARING:
Plan to Share IPD: Undecided